CLINICAL TRIAL: NCT05876156
Title: Immersive Virtual Reality for Enhancement of Physical Activity in Pediatric Oncology : a Randomised Control Study (iMOVE)
Brief Title: iMOVE: Virtual Reality PT Versus Traditional PT
Acronym: iMOVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-70481
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Physical Health
Keywords: Virtual Reality; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VRPT then Traditional PT (Experimental): Participants will receive Virtual Reality assisted Physical Therapy sessions (VRPT) in the first Physical Therapy (PT) session and will receive traditional Physical Therapy sessions (standard care) in the second Physical Therapy session under the supervision of the accredited physical therapist.
  Interventions: Behavioral: Virtual Reality Physical Therapy; Behavioral: Traditional Physical Therapy
- Traditional PT then VRPT (Experimental): Participants will receive traditional Physical Therapy (PT) sessions (standard care) in the first Physical Therapy session and Virtual Reality assisted Physical Therapy sessions (VRPT) in the second Physical Therapy session under the supervision of the accredited physical therapist.
  Interventions: Behavioral: Virtual Reality Physical Therapy; Behavioral: Traditional Physical Therapy

INTERVENTIONS:
Behavioral: Virtual Reality Physical Therapy — Participants are allowed to freely choose one game from the game list. Participant will be asked to wear a validated activity tracker - ActiGraph. Baseline heart rate will be collected for 1 minute. Participants will be wearing the ActiGraph during Physical Therapy session. Participants receiving VR intervention will be instructed to wear an Oculus Quest 2 headset (Meta, Inc., Menlo Park, CA) and participate in VR applications under the supervision of the physical therapist.
  Other Names: VRPT
Behavioral: Traditional Physical Therapy — Participants will receive traditional Physical Therapy sessions (standard care) under the supervision of the accredited physical therapist. Participants will be wearing the Actigraph during Physical Therapy session. Participants will perform regular physical exercise, such as 20 minutes walking or biking on a stationary bike, under the supervision of a physical therapist.

SUMMARY:
This pragmatic, crossover, randomized controlled study evaluates the efficacy of virtual reality assisted physical therapy (VRPT) for improving the physical activity of hospitalized children as compared to traditional physical therapy. This is a pilot study that will be used to identify patient populations that can benefit the most from VRPT and estimate this effect for future studies.

Patients with a significant neurological condition, major developmental disability, active infection of the face or hand, history of severe motion sickness, history of seizures caused by flashing light or had a major surgery within the last 48 hours will be excluded.

DETAILED DESCRIPTION:
Childhood cancer is a significant health concern worldwide. Despite improved 5-year survival rates (80%-85%), children undergoing treatment face physiological and psychosocial challenges, including chronic pain, limited mobility, muscle loss, low bone density, and mental distress. To mitigate negative therapy-related adverse health outcomes and improve quality of life, supportive care measures are emphasized during cancer treatments. The US Department of Health & Human Services advises Pediatric oncology patients to engage in 30 minutes of moderate-intensity physical activity, 3 times a week, for a healthy lifestyle. Regular exercise during and after treatment profoundly impacts a child's physical, psychological, and social well-being. Inpatient and outpatient physical therapy is commonly suggested for patients. Yet, traditional physical therapy is usually monotonous and repetitive, leading to boredom and decreased adherence. Limited exercise variation may fail to captivate attention and provide motivation for consistent participation.

Virtual reality physical therapy (VRPT) provides dynamic and interactive exercise, overcoming traditional therapy's boredom. Exergaming offers fun and excitement through engaging virtual environments and gameplay. It enhances motivation, sustains interest, and encourages longer exercise. Personalized and adaptive interventions in virtual reality target individual needs and allow progress tracking.

ELIGIBILITY:
Inclusion Criteria:

* Between age 10-25 years
* Diagnosed with cancer
* Has an active physical therapy consultation
* Anticipated inpatient stay for at least 3-days with the second PT session following between 24-72 hours after the first PT session
* Ability to understand and the willingness to personally sign the written Institutional Review Board (IRB) approved informed consent document by Legally Authorized Representative (LAR) if participant <18 years old or by participant if 18+
* Ability to understand and the willingness to personally sign the written IRB approved informed assent document for patient <18 years old.

Exclusion Criteria:

* Legal guardian does not present to obtain consent.
* Child with a significant neurological condition, or major developmental disability.
* Child with active infection of the face or hand.
* A history of severe motion sickness.
* A history of seizures caused by flashing light.
* Major surgery within the last 48 hours.
* Does not speak English (required for surveys)
* With visual impairments or any degree of developmental delays
* Child on mechanical ventilation or ventilatory support

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
ActiGraph data points | During physical therapy session
  Compare the total Metabolic Equivalent of Task (METs) rate of pediatric oncology patients when undergo virtual reality assisted physical therapy and traditional physical therapy measured by ActiGraph watch

SECONDARY OUTCOMES:
Total exercise time spend in moderate-vigorous activity | During physical therapy session
  Compare the difference in total exercise time in moderate-vigorous activity of pediatric oncology patients when undergo virtual reality assisted physical therapy and traditional physical therapy measured by ActiGraph watch
Total exercise time spend in sedentary activity | During physical therapy session
  change in total exercise time in sedentary activity of pediatric oncology patients when undergoing virtual reality assisted physical therapy compared to traditional physical therapy measured by ActiGraph watch. For this measure, both absolute change and difference in the proportion of time spent will be evaluated.
Total exercise time spend in light activity | During physical therapy session
  change in the total exercise time in light activity of pediatric oncology patients when undergoing virtual reality assisted physical therapy compared to traditional physical therapy measured by ActiGraph watch. For this measure, both absolute change and difference in the proportion of time spent will be evaluated.
Change in OMNI RPE survey scores | immediately after the physical therapy session
  Patients will self-report fatigue according to the Adult OMNI-Walk/Run RPE Scale (OMNI RPE) scale after both the VR and standard of care portion. The OMNI RPE is an 11-categories perceived exertion rating scale with a numerical rating from 0 to 10 (0= Not Tired at All, 10= Very, Very Tired).
Feasibility and Usability Survey (Parent) | immediately after the physical therapy session
  Tabulate the self -formulated Feasibility and Usability Survey. This questionnaire consists of 12 items, including 5 Likert questions, 6 yes/no questions and 1 open-end question. Measures are to be graded using a 1-10 scale, from 1=not at all, to 10=very much.
Acceptability of Intervention Measure (AIM) survey | immediately after the physical therapy session
  This questionnaire consists of 4 items. Measures are to be graded using a 1-5 scale, from 1=completely disagree, to 5= completely agree
Intervention Appropriateness Measure (IAM) survey | immediately after the physical therapy session
  This questionnaire consists of 4 items. Measures are to be graded using a 1-5 scale, from 1=completely disagree, to 5= completely agree
Feasibility of Intervention Measure (FIM) survey | immediately after the physical therapy session
  This questionnaire consists of 4 items. Measures are to be graded using a 1-5 scale, from 1=completely disagree, to 5= completely agree

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Caruso, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Childrens Hospital Stanford, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No